CLINICAL TRIAL: NCT01503541
Title: The Development of Predictive Biomarker Models for Patients Receiving Standard Induction Chemotherapy With and Without Gemtuzumab Ozogamicin
Brief Title: S9031-9333-0106-0112-A Study of Biomarkers in Samples From Patients With Acute Myeloid Leukemia Treated With Standard Chemotherapy With or Without Gemtuzumab Ozogamicin
Status: Completed | Type: Observational
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: S9031-9333-0106-0112-A; S9031-9333-0106-0112-A (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2012-01-01; First posted 2012-01-04 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2014-01

CONDITIONS: Leukemia
Keywords: adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with del(5q); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Congenital Abnormalities; Leukemia, Myeloid, Acute | interventions — Gene Expression Profiling; Polymerase Chain Reaction

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Genetic: DNA analysis
Genetic: RNA analysis
Genetic: gene expression analysis
Genetic: mutation analysis
Genetic: polymerase chain reaction
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of bone marrow and blood from patients with cancer in the laboratory may help doctors identify and learn more about biomarkers related to cancer.

PURPOSE: This research trial studies biomarkers in samples from patients with acute myeloid leukemia treated with standard chemotherapy with or without gemtuzumab ozogamicin.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine whether measuring biomarkers in less-differentiated acute myeloid leukemia (AML) blasts significantly improves their predictive accuracy to predict clinical outcomes for patients receiving induction/consolidation chemotherapy with and without gemtuzumab ozogamicin.
* To develop and validate novel predictive biomarker models for predicting clinical outcomes for AML patients receiving induction/consolidation chemotherapy with and without gemtuzumab ozogamicin.

OUTLINE: DNA and RNA extracted from archived bone marrow and peripheral blood samples are analyzed for genomic mutations (CEBPA, FLT3, IDH1/2, KIT, NPM1, RUNX1, TP53, and WT1) and transcriptional biomarkers (BAALC, CCNA1, CD34, CEBPA, ERG, EVI1, FLT3, IL3RA, MCL1 [two splice variants], MN1, RUNX1, and WT1) by PCR and real-time PCR. Data are then analyzed by the Gene Scan software.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pretreatment bone marrow (BM) and peripheral blood (PB) samples obtained from Southwest Oncology Group ( SWOG) Leukemia Repository for adult patients enrolled on SWOG-9031, SWOG-9333, SWOG-S0106, and SWOG-S0112
* Samples restricted to those patients from these studies with at least 3 or more vials of remaining material in the SWOG Leukemia Repository and vials containing at least 1.5 x 10^7 cells/vial
* Samples from patients who received standard induction with cytarabine (ARA)/daunorubicin hydrochloride (DNR) with the addition of gemtuzumab ozogamicin (Mylotarg®) on one arm of S0106

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Specimens from patients consenting to future research on S9031, S9333, S0106 and S0112
Sampling Method: Non-Probability Sample
Enrollment: 365 (Actual)
Dates: Start 2011-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Biomarker assays in highly purified populations of AML myeloblasts are more predictive of clinical outcomes as compared to the same tests examining unsorted cells | immediate
Development of risk-assessment biomarker model for clinical outcomes | immediate

CONTACTS AND LOCATIONS:
Overall Officials: Derek L. Stirewalt, MD, Principal Investigator — Fred Hutchinson Cancer Center